CLINICAL TRIAL: NCT01272596
Title: Evaluation of Low Contrast Sloan Visual Charts as Method for the Assessment of Disease Progression in Multiple Sclerosis
Brief Title: Evaluation of Sloan-Charts for Assessment of Disease Progress in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis Germany GmbH (Unknown)
Responsible Party: Principal Investigator, Jan-Markus Dörr, PI, Charite University, Berlin, Germany
Other Study IDs: Sloan-Study
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Visual Contrast Acuity; Visual Contrast Sensitivity; Sloan Charts
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Patients: Patients with Clinically Isolated Syndrome or definite Multiple Sclerosis (either relapsing-remitting or secondary progressive)

SUMMARY:
Impairment of visual deficits, in particular contrast acuity and contrast impairment are frequent symptoms in MS. However, visual function is not appropriately covered by the standard tools for clinical assessment, namely, the EDSS and the MSFC.

The primary aim of this study is to investigate, whether in MS patients contrast acuity and sensitivity change over a period of two years.

Secondary aims are the correlation of visual contrast parameters with structural retinal changes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Isolated Syndrome or definite MS (relapsing-remitting or secondary progressive course)
* Written Informed Consent

Exclusion Criteria:

* Relapse within the last 30 Days
* Significant Cognitive Impairment
* Severely Decreased Visual Acuity
* Preexisting Severe Retinal Pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Clinically Isolated Syndrome or Definite Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Visual Contrast Acuity | 24 Months

SECONDARY OUTCOMES:
Structural and Functional Changes of Optic Pathway | 24 Months
Clinical Neurological Assessment | 24 Months
Quality of Life | 24 Months
Contrast Sensitivity | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Dörr, MD, Principal Investigator — NeuroCure Clinical Research Center, Charité Universitaetsmedizin Berlin
Locations (1):
- NeuroCure Clinical Reserach Center, Charité Universitaetsmedizin, Berlin, Germany

REFERENCES:
- See also: NeuroCure Clinical Research Center, Charité Berlin, Germany — https://neurocure.de/ncrc/ueber-uns.html